CLINICAL TRIAL: NCT06726018
Title: Exploring Pain Modulation Mechanisms: A Study of TMS and Repeated Conditioned Pain Modulation
Brief Title: Exploring Pain Modulation With TMS and Repeated Pain Conditioning in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Priyanka Rana, PT, MPT, PhD (Other)
Responsible Party: Sponsor-Investigator, Priyanka Rana, PT, MPT, PhD, Assistant Professor, University of Texas, El Paso
Organization: University of Texas, El Paso (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2261897-1
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult
Keywords: Pain; Pain Modulation; Conditioned Pain Modulation; Transcranial Magnetic Stimulation; Chronic Pain Mechanisms
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Exposure (HE) (Experimental): Participants will receive five sessions total: four sessions of the Intervention, CPM and TMS as an outcome in every session and questionnaires and QST as an outcome in the first and fifth sessions.
  Interventions: Behavioral: Conditioned Pain Modulation (CPM)
- Low Exposure (LE) (Active Comparator): Participants will receive only two sessions in total: one session of the intervention, questionnaires, quantitative sensory testing, CPM and TMS as an outcome at both sessions.
  Interventions: Behavioral: Conditioned Pain Modulation (CPM)
- No Exposure (NE) (No Intervention): Participants will receive only two sessions in total: questionnaires, quantitative sensory testing, and TMS as an outcome at both sessions.

INTERVENTIONS:
Behavioral: Conditioned Pain Modulation (CPM) — Participants will receive a testing stimulus of pressure applied per ascending intensity at the web space of the foot until the pain reaches 40 out of 100, then discontinued. After testing the stimulus, participants will then receive a conditioning stimulus by immersing the non-dominant hand into the water-cooled by refrigeration unit with a temperature of 6 degree Celsius (males) or 8 degree Celsius (females) for 60 seconds. Subjects will be asked to rate the cold pain during the four 60-second trials. Participants completely removed their hand from the cold pressor for 30 seconds following each of the four 60-second immersions, during which time the testing stimulus will be re-applied per the sequential paradigm to the web space of the foot. Participants complete four 60-second periods of immersion.
  Arms: High Exposure (HE); Low Exposure (LE)

SUMMARY:
Conditioned pain modulation (CPM) is the behavioral measure of diffuse noxious inhibitory control (DNIC), an endogenous pain inhibitory pathway in which pain inhibits pain. CPM is less efficient in individuals with chronic pain conditions, and it is a predictor for the development of chronic pain. Continuous stimulation of central/cortical mechanisms through engaging CPM might alter pain processing and improve pain inhibition. Transcranial Magnetic Stimulation (TMS) is a valuable tool for assessing how effectively the brain's central and cortical mechanisms engage in pain inhibition, particularly through pathways like CPM.

While alterations in cortical excitability related to analgesic-induced pain inhibition have been documented, the effects of continuous stimulation of central pain pathways, along with the mediating influence of psychosocial factors, remain underexplored. This study aims to investigate the central pain modulatory mechanisms, as assessed by CPM, and cortical excitability, as measured by TMS, in healthy participants. Additionally, the study will evaluate the impact of sociocultural factors, including ethnic identity, optimism, resilience, perceived stress, and marginalization, on the magnitude and efficiency of CPM responses.

The successful completion of this research will determine how cortical excitability changes due to training and whether these changes are mediated by psychosocial factors.

DETAILED DESCRIPTION:
Background:

Pain and Its Burden

Pain is a prevalent and complex health condition that significantly impacts individuals, families, and society as a whole. Of the 39.4 million adults experiencing pain most days and persisting for over three months, nearly two-thirds report it as "constantly present," with over half describing it as "unbearable and excruciating" . Pain can be categorized into physiological and pathological types. Nociceptive and inflammatory pain are physiological responses that serve protective and adaptive functions, whereas pathological pain is considered non-protective and maladaptive.

Central Mechanisms in Pain Modulation

Laboratory-based quantitative sensory testing (QST) evaluates sensory function using psychophysical methods, teasing out components of the nervous system that demonstrate loss or gain of sensory function contributing to pain. The conditioned pain modulation (CPM) paradigm is a dynamic QST measure of a pain inhibitory process in which pain sensitivity in one area decreased in response to a remotely applied painful stimulus and is used to assess the ability of the person to endogenously inhibit pain. CPM may be a valuable tool in directing mechanistic-based approaches for treating painful conditions. For example, individuals with painful diabetic neuropathy and poorly functioning CPM have more significant analgesia when given duloxetine, a medication that augments conditioned pain modulation. Additionally, identifying and treating the source of pain is associated with positive changes in CPM. Healthy individuals demonstrate more efficient CPM when compared with people in pain and a systematic review of adults with chronic pain revealed that CPM efficiency improves after a reduction in clinical pain. For example, total hip arthroplasty for treating painful osteoarthritis reduces joint pain and improves post-operative CPM. Collectively, these studies suggest that the CPM test has the potential to predict risk and treatment outcomes for chronic pain, therefore CPM may be considered an essential treatment moderator and mediator.

The activation of central mechanisms, particularly endogenous inhibitory systems, is proposed as a fundamental process underlying various pain management interventions. Descending pain inhibitory systems, which are part of central mechanisms, play a crucial role in mediating the analgesic effects of interventions such as manual therapy. Manual therapy stimulates afferent neuronal inputs that activate the central nervous system's descending pathways to inhibit pain. Conditioned Pain Modulation (CPM) shares a similar mechanism, inhibiting pain through descending modulation pathways. Continuous stimulation of these central mechanisms through CPM could potentially alter pain processing and enhance pain inhibition.

Role of Transcranial Magnetic Stimulation (TMS) in Pain Inhibition

TMS is a non-invasive neurophysiological technique that employs magnetic fields to modulate and measure brain activity. It is particularly valuable in studying pain inhibition mechanisms and understanding brain processing of pain stimuli. TMS measures cortical excitability by delivering magnetic pulses to specific brain regions and recording motor-evoked potentials. This technique is increasingly used to investigate neural mechanisms involved in pain perception and inhibition, especially in conditions where these processes may be disrupted, such as chronic pain disorders. By targeting regions like the primary motor cortex or prefrontal cortex, TMS helps researchers examine the roles of excitatory and inhibitory pathways in pain suppression or facilitation.

TMS and Conditioned Pain Modulation (CPM)

TMS is employed to assess the brain's natural ability to inhibit pain through CPM paradigms. In these studies, TMS is used to evaluate how effectively a person's brain can inhibit pain when a secondary, often painful, stimulus is introduced. Individuals with lower cortical excitability in response to noxious stimuli are thought to have stronger endogenous pain inhibition, whereas those with higher cortical excitability may have impaired pain inhibition mechanisms.

Integrating TMS and CPM in Pain Research

In this study, the investigators will employ CPM as both an assessment tool and an intervention method. Combining TMS and CPM provides a comprehensive approach to understanding the neurophysiological and psychosocial factors influencing pain modulation. TMS offers direct measurements of cortical excitability, while CPM assesses an individual's ability to modulate pain through endogenous pathways. As an intervention, CPM will be utilized to potentially modulate nervous system responses. This approach aims to enhance pain inhibitory mechanisms through repeated exposure to controlled painful stimuli, potentially leading to adaptive neuroplastic changes. By simultaneously examining cortical excitability via TMS and endogenous pain modulation through CPM, the investigators aim to delineate the complex interplay betthe investigatorsen central and peripheral mechanisms underlying pain processing.

Research Gaps and Future Directions

Research has demonstrated alterations in cortical excitability associated with pain experiences, predominantly focusing on chronic pain conditions. However, there is a paucity of investigations examining cortical excitability in the context of experimental pain responses and modifications in central pain processing mechanisms. Moreover, although psychological factors such as catastrophizing and hypervigilance have been associated with pain sensitivity, the role of sociocultural constructs such as ethnic identity, optimism, resilience, perceived stress, marginalization, and their relationship with pain inhibition and cortical excitability via continuous stimulation of central mechanisms remains underexplored.

Specific Aims:

Aim 1: To investigate the effect of repeated CPM exposure on cortical excitability Hypothesis 1: Repeated CPM exposure will be associated with alterations in cortical excitability.

Aim 2: To investigate the mediation effect of sociocultural factors on the relationship between repeated CPM exposure and cortical excitability.

Hypothesis 2: Sociocultural factors will mediate the relationship between repeated CPM exposure and cortical excitability, influencing the degree of cortical excitability changes.

Aim 3: To investigate the mediation effect of sociocultural factors on the relationship between repeated CPM exposure and pain sensitivity.

Hypothesis 3: Sociocultural factors will mediate the relationship between repeated CPM exposure and pain perception.

Impact and Significance

This investigation into pain inhibitory mechanisms has the potential to significantly advance our understanding of chronic pain pathophysiology and identify novel therapeutic targets. By elucidating the neurobiological processes underlying pain perception and modulation, this study addresses critical clinical questions regarding changes in cortical excitability and the influence of psychosocial factors on pain perception following nervous system training. The primary innovation of this proposal lies in its comprehensive assessment of central pain mechanisms through transcranial magnetic stimulation (TMS) in conjunction with continuous stimulation via Conditioned Pain Modulation (CPM). This approach, combined with the evaluation of sociocultural constructs such as ethnic identity, optimism, resilience, and marginalization among Hispanic and non-Hispanic populations, offers a unique perspective on pain processing.

By bridging the gap between neurophysiological mechanisms and sociocultural influences on pain, this research has the potential to significantly impact both our theoretical understanding of chronic pain and clinical practice in pain management. The insights gained could inform more targeted and effective interventions, ultimately improving the quality of life for individuals suffering from chronic pain.

Research Plan:

The study in this proposal will be based on psychophysical data and self-reported questionnaires using methods approved by the University of Texas El Paso Institutional Review Board. This prospective experimental study involves healthy participants who will undergo baseline assessments, including psychological questionnaires and psychophysical approaches to measuring individual sensitivity, endogenous pain modulation and transcranial magnetic stimulation. Immediately after an intervention period, participants will be reassessed. All assessments will be performed by an evaluator who will be blind to psychological measure data and group assignment.

Participants:

Seventy individuals will be recruited by posted fliers approved by the IRB on the University of Texas El Paso campus and the El Paso community.

Inclusion criteria: a) pain-free; b) between 18-75 years old. Exclusion criteria: Participants will not be excluded based on race or gender but will be excluded if they meet any of the following a) non-English speaking; b) systemic medical condition is known to affect sensation; c) regular use of prescription pain medication to manage pain; d) current or history of chronic pain condition; e) currently using blood thinning medication; f) any blood clotting disorder such as hemophilia; g) any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise; h) involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling.

Individuals meeting the preliminary screening criteria will undergo an in-person TMS safety screen (English and Spanish language versions included in study case report forms). Briefly, individuals will pass the TMS safety screen if they have no metal in the head or eyes, no pacemakers, shunts, or lines, no history of craniotomy, no history of focal seizures. A detailed screening questionnaire is included in the submitted case report forms.

Recruitment and Informed Consent Procedure:

Potential participants for this study will be recruited through a comprehensive strategy employing multiple channels. Recruitment methods will include strategically placed flyers, targeted social media campaigns, word-of-mouth referrals, and direct recommendations from healthcare providers. Individuals expressing interest in the study will be encouraged to contact the research team directly. The primary Investigator or co-investigator will read from an IRB-approved phone script or respond through an IRB-approved e-mail script to provide an overview of basic information about the study and answer questions. Participants wishing to participate will be scheduled for the formal consent process with either the Principal Investigator or co-investigator. Informed consent will occur in the Department of Physical Therapy lab space at UTEP. At that time, the primary Investigator or co-investigator will explain the study procedure, study purpose, benefits/risks of participating, and use of protected health information. The investigators will ensure appropriate time is spent with the participant to answer any questions and ensure he or she understands the procedures and risks associated with the study. If the participant chooses to participate, informed consent will be obtained from the participant as appropriate.

Measures:

Measures will be collected by the primary investigator, co-investigator, and/or research assistant under the direct supervision of the primary or co-investigator.

Questionnaires:

Demographic and Historical Factors: Study participants will complete a standard intake information form including gender, age, employment status, marital status, educational level, and health history.

The Brief Pain Inventory - Short Form (BPI-sf): The Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a pain and the impact of this pain on daily functioning. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as participants can imagine, and contributes with the same weight to the final score, ranging from 0 to 40.

The Multigroup Ethnic Identity Measure (MEIM): The MEIM is a 15-item scale that measures ethnic identity. The items are rated on a four-point Likert scale, with 1 indicating "strongly disagree" and 4 indicating "strongly agree". Higher scores indicating a stronger ethnic identity.

Life Orientation Test-Revised (LOT-R): The LOT-R is a 10-item self-report scale that measures how optimistic or pessimistic a person feels about the future. It measures trait optimism. The LOT-R uses a 5-point Likert scale, with 0 meaning "strongly disagree" and 4 meaning "strongly agree". Items are summed, yielding a range from 0 to 32 and Higher scores indicate greater levels of optimism.

State Optimism Measure (SOM): The SOM is a 7-item measure that measures a person's state of optimism. It scored from 1 to 7 and higher scores indicate with a higher score indicating greater state optimism. It has been shown to be reliable and valid in both general and clinical populations.

Brief Resilience Scale (BRS): The BRS is a test that measures a person's ability to recover from stress. It's made up of six items that are rated on a five-point scale, with half of the items being positively worded and half negatively worded. Higher average scores indicate higher levels of perceived resilience. Three items are reverse-coded before scoring.

The Perceived Societal Marginalization (PSM): The PSM scale is a tool that measures how people perceive their social group's lack of recognition and insignificance in the areas of culture, politics, and the economy. The scale's items are scored on a 6-point Likert scale, with 1 representing "strongly disagree" and 6 representing "strongly agree". A higher total score indicates a higher level of perceived societal marginalization.

Anxiety about Pain Testing: A single item visual analogue scale (VAS) for Anxiety about Pain Testing was administered before every session of the protocol. The VAS was 100mm long and participants were instructed that the anchors were "no anxiety about pain testing" on the left and "worst anxiety about pain testing imaginable" on the right.

Pain Catastrophizing Scale (PCS): The Pain Catastrophizing Scale is a 13-item questionnaire in which individuals respond to a statement on a five-point ordinal scale from 0 to 4. Individuals respond to the question in terms of a prior painful episode, and higher scores indicate higher pain catastrophizing levels.

Perceived Stress Scale (PSS): The PSS is a 14-item measure that measures a person's perception of stress. It scored from 0 to 56 and higher scores indicate with a higher score indicating more stress. It has been shown to be reliable and valid in both general and clinical populations.

Quantitative Sensory Testing:

Participants will complete Quantitative Sensory Testing (QST). The researcher will record pain responses to the quantitative sensory testing protocol using the numeric pain rating scale (NRS). The numeric pain rating scale is a 100-point scale in which patients verbally rate their pain from 0, indicating "no pain," to 100, indicating "the most intense pain sensation imaginable." The NRS demonstrates sound psychometric properties.

Slow Ramp: A slowly ramping thermal stimulus will be delivered to the skin of the participant's dominant forearm using a computer controlled TSAII NeuroSensory Analyzer from Medoc, Inc. Thermal stimuli will increase from a baseline of 35 degrees Celsius to a maximum of 51 degree Celsius in ascending one-degree intervals, each stimulus presented for 1-sec. Participants will be instructed to indicate when the sensation first changes from warmth to pain (pain threshold) and when the sensation becomes "so painful participants can no longer tolerate it" (pain tolerance). This procedure will be repeated two times with a pseudorandom interval 1-sec/min and the average temperature to achieve the threshold and tolerance analyzed.

After sensations: The participants will be asked to rate the magnitude of their pain sensation following the removal of the thermode. The research assistant will cue the participants to rate their pain every 10 seconds. These ratings will be obtained for 60 seconds. These response ratings are also primarily C-fiber mediated.

Pressure Pain Threshold: An algometer with a 1 cm diameter rubber tip will be applied at 1 kg/s to the dominant hand at the first dorsal interosseous muscle. Participants will be instructed to indicate when the sensation first changes from pressure to pain (pain threshold). This procedure will be repeated two times, and the average pressure to threshold will be analyzed.

Conditioned Pain Modulation (as an assessment): Participants will receive a testing stimulus of pressure applied to the web space of the dominant foot (the foot that participant instinctively kick). Pressure will be applied per ascending intensity until the pain reaches 40 out of 100, then discontinued. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when participants feel pain equal to 40 out of 100." This will be repeated two times, and the average will be analyzed (Yarnitsky et al., 2015). Participants will then receive a conditioning stimulus contact heat stimulus applied to the thenar of the non-dominant hand and non-dominant forearm for 60 s at an intensity of 46.5 ◦C (Matre, 2013). Subjects will be asked to rate the heat pain and unpleasantness during a 60-second trial. Subjects will be instructed that they may remove their hand at any time if the heat is intolerable. After 60 seconds, the contact heat will be completely removed, and the testing stimulus will be re-applied to the web space of the dominant foot. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation (Yarnitsky et al., 2012).

TMS testing: Individuals meeting the TMS safety criteria will undergo baseline TMS to determine the resting motor threshold, short-interval intracortical inhibition (SICI) protocols. Both are established, reliable, valid protocols to measure motor cortical excitability and inhibition, respectively. TMS will be delivered using a D702 coil connected to Magstim 2002 magnetic stimulators via a Bistim unit (Magstim, UK). A resting motor threshold, defined as the stimulus intensity required to elicit a 50uV motor evoked potential in 5 out of ten TMS stimuli at the motor hotspot for dominant abductor pollicis brevis (APB) muscle will be determined with the participant seated, both shoulders in neutral, forearm supinated, and palms resting on a pillow in their lap. Twenty pulses of 1mV peak to peak motor evoked potentials will be recorded to assess cortical excitability. SICI will be investigated by applying a subthreshold conditioning stimulus before the test stimulus using a 1ms (SICI1ms) or a 3ms (SICI3ms) interstimulus interval to assess the two SICI phases considered to reflect extrasynaptic and synaptic GABAA receptor activity respectively. SICI will be obtained with conditioning stimulus intensities of 50, 65, 80, and 95% of the AMT and a test stimulus of 1mV amplitude. In addition, short-interval intracortical facilitation (SICF) will similarly be determined using a 10-15ms interval with conditioning stimulus intensities same as SICI. Similar TMS procedures are currently being used in the Geed Lab for a UTEP-IRB approved protocol (#2076486-1, Neuroplasticity and hand function recovery after stroke). The investigators expect to record 20 motor evoked potential (MEP) pulses, 20 SICI, and 20 SICF pulses in each participation before and after the CPM intervention.

Procedure:

Participants who consent will sign up for individual blocks of testing time (90 minutes) to take part in the experiment. Participants will be asked to complete the Ethical Identity, BPI, LOT-R, SOM, BRS, PSM and PSS questionnaires before and after the protocol. Participants will complete VAS for Anxiety about Pain Testing before every protocol session. Blood pressure will be assessed with a digital blood pressure monitor before every session. If blood pressure exceeds 140/90 mmHg, the participant will be removed from the study session and notified of the blood pressure reading. Next, TMS, CPM and a baseline assessment of pain sensitivity will be completed. After testing, participants sit quietly for 15 minutes to allow changes in pain sensitivity to normalize after pre-intervention CPM testing (Lewis et al., 2012). Healthy participants will be randomized to one of three groups: High Exposure (HE), Low Exposure (NE) and No Exposure (NE).

High Exposure: Participants will receive five sessions total: four sessions of the Intervention, CPM and TMS as an outcome in every session and questionnaires and QST as an outcome in the first and fifth sessions.

Low Exposure: Participants will receive only two sessions in total: one session of the intervention, questionnaires, quantitative sensory testing, CPM and TMS as an outcome at both sessions.

No Exposure: Participants will receive only two sessions in total: questionnaires, quantitative sensory testing, and TMS as an outcome at both sessions.

High exposure group will be attending 5 sessions (about once every 72 hours) for two weeks. The Low Exposure and No Exposure group come twice (the second visit about 2 weeks later). Visits can last 2.5 to 3 hours.

Intervention:

CPM: Participants will receive a testing stimulus of pressure applied to the web space of the dominant foot. Pressure is applied per ascending intensity until the pain reaches 40 out of 100, then discontinued. Participants will be instructed to say "stop" or "pain" so the stimulus can be terminated "when participants feel pain equal to 40 out of 100." This will be repeated twice, and the average will be analyzed (Yarnitsky et al., 2015). Participants will then receive a conditioning stimulus by immersing non-dominant hand into the water cooled by a refrigeration unit (NESLAB RTE 7 Digital One, Thermo Scientific Co., Massachusetts, USA) that circulates water continuously to maintain a constant temperature of six degree Celsius (males) or eight degree Celsius (females) for 60 seconds. Subjects will be asked to rate the cold pain and unpleasantness during the four 60-second trials. Subjects will be instructed that they may remove their hand at any time if the water is intolerable. If this occurs, or if subjects rate the pain higher than 50 (0-100 scale), the bath temperature will be increased for the subsequent trial. If the ratings are less than 20, a small amount of ice was added to lower the temperature by up to 4o Celsius. Participants completely removed their hand from the cold pressor for 30 seconds following each of the four 60-second immersions, during which time the testing stimulus will be re-applied per the sequential paradigm to the web space of the foot. Participants complete four 60-second periods of immersion. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation.

Immediately following the assigned intervention, TMS and measures will be re-assessed as described above.

ELIGIBILITY:
Inclusion Criteria:

* pain-free
* between 18-75 years old.

Exclusion Criteria:

Participants will not be excluded based on race or gender but will be excluded if they meet any of the following:

* non-English speaking
* systemic medical condition is known to affect sensation
* regular use of prescription pain medication to manage pain
* current or history of chronic pain condition
* currently using blood thinning medication
* any blood clotting disorder such as hemophilia
* any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise
* involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling
* metal in the head or eyes, pacemakers, shunts, or lines, history of craniotomy, history of focal seizures
* Migraine and persistent headaches.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Conditioned Pain Modulation as an assessment | Two-weeks
  Participants will receive a testing stimulus of pressure applied per ascending intensity at the web space of the foot until the pain reaches 40 out of 100, then discontinued. After testing the stimulus, Participants will receive a conditioning stimulus contact heat stimulus applied to the thenar of the left hand for 60 s at an intensity of 46.5 ◦C. Subjects will be asked to rate the heat pain during the four 60-second trials. Subjects will be instructed that they may remove their hand at any time if the heat is intolerable. After 60 seconds, the contact heat will be completely removed, and the testing stimulus will be re-applied to the web space of the dominant foot. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation
Transcranial Magnetic Stimulation | Two-weeks
  Individuals meeting the TMS safety criteria will undergo baseline TMS to determine the resting motor threshold, short-interval intracortical inhibition (SICI) protocols. Both are established, reliable, valid protocols to measure motor cortical excitability and inhibition, respectively. TMS will be delivered using a D702 coil connected to Magstim 2002 magnetic stimulators via a Bistim unit (Magstim, UK). A resting motor threshold, defined as the stimulus intensity required to elicit a 50uV motor evoked potential in 5 out of ten TMS stimuli at the motor hotspot for dominant abductor pollicis brevis (APB) muscle will be determined with the participant seated, both shoulders in neutral, forearm supinated, and palms resting on a pillow in their lap. Twenty pulses of 1mV peak to peak motor evoked potentials will be recorded to assess cortical excitability. SICI will be investigated by applying a subthreshold conditioning stimulus before the test stimulus using a 1ms (SICI1ms) or a 3ms (SICI
Quantitative Sensory Testing | Two-weeks
  Slow Ramp Protocol: A computer-controlled TSAII NeuroSensory Analyzer (Medoc, Inc.) will deliver a thermal stimulus to the dominant forearm, starting at 35°C and increasing to 51°C in 1°C increments, each lasting 1 seconds. Participants will report when the sensation changes from warmth to pain (pain threshold) and when it becomes intolerable (pain tolerance). The procedure will be repeated twice with a pseudorandom interval (1 sec/min), and average thresholds and tolerances will be analyzed.
  Post-Stimulus Ratings: Participants will rate pain every 10 seconds for 60 seconds after the thermode is removed. These ratings primarily reflect C-fiber-mediated responses.
  Pressure Pain Threshold: Using an algometer with a 1 cm rubber tip, pressure will be applied at 1 kg/s to the first dorsal interosseous muscle of the dominant hand. Participants will report when the sensation changes from pressure to pain (pain threshold). The procedure will be repeated twice. Average will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Movement Science, University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein MM, Treister R, Raij T, Pascual-Leone A, Park L, Nurmikko T, Lenz F, Lefaucheur JP, Lang M, Hallett M, Fox M, Cudkowicz M, Costello A, Carr DB, Ayache SS, Oaklander AL. Transcranial magnetic stimulation of the brain: guidelines for pain treatment research. Pain. 2015 Sep;156(9):1601-1614. doi: 10.1097/j.pain.0000000000000210. PMID 25919472
- [Background] Kennedy J, Roll JM, Schraudner T, Murphy S, McPherson S. Prevalence of persistent pain in the U.S. adult population: new data from the 2010 national health interview survey. J Pain. 2014 Oct;15(10):979-84. doi: 10.1016/j.jpain.2014.05.009. PMID 25267013
- [Background] Ibancos-Losada MDR, Osuna-Perez MC, Castellote-Caballero MY, Diaz-Fernandez A. Conditioned Pain Modulation Effectiveness: An Experimental Study Comparing Test Paradigms and Analyzing Potential Predictors in a Healthy Population. Brain Sci. 2020 Aug 30;10(9):599. doi: 10.3390/brainsci10090599. PMID 32872642
- [Background] Hinz A, Sander C, Glaesmer H, Brahler E, Zenger M, Hilbert A, Kocalevent RD. Optimism and pessimism in the general population: Psychometric properties of the Life Orientation Test (LOT-R). Int J Clin Health Psychol. 2017 May-Aug;17(2):161-170. doi: 10.1016/j.ijchp.2017.02.003. Epub 2017 Mar 31. PMID 30487891
- [Background] Harris KM, Gaffey AE, Schwartz JE, Krantz DS, Burg MM. The Perceived Stress Scale as a Measure of Stress: Decomposing Score Variance in Longitudinal Behavioral Medicine Studies. Ann Behav Med. 2023 Sep 13;57(10):846-854. doi: 10.1093/abm/kaad015. PMID 37084792
- [Background] Goubert D, Danneels L, Cagnie B, Van Oosterwijck J, Kolba K, Noyez H, Meeus M. Effect of Pain Induction or Pain Reduction on Conditioned Pain Modulation in Adults: A Systematic Review. Pain Pract. 2015 Nov;15(8):765-77. doi: 10.1111/papr.12241. Epub 2014 Nov 11. PMID 25387406
- [Background] Fong A, Schug SA. Pathophysiology of pain: a practical primer. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):8S-14S. doi: 10.1097/PRS.0000000000000682. PMID 25255013
- [Background] Bellei-Rodriguez CE, Colloca L, Lorrain D, Marchand S, Leonard G. Nocebo Effect on Pain Perception and Attention with Children With and Without Attention Deficit And/Or Hyperactivity Disorder. J Dev Behav Pediatr. 2024 Nov-Dec 01;45(6):e537-e544. doi: 10.1097/DBP.0000000000001314. Epub 2024 Nov 11. PMID 39377730
- [Background] 6. Chowdhury, N. S., Chiang, A. K., Millard, S. K., Skippen, P., Chang, W.-J., Seminowicz, D. A., & Schabrun, S. M. (2023). Alterations in cortical excitability during pain: A combined TMS-EEG Study. BioRxiv : The Preprint Server for Biology. https://doi.org/10.1101/2023.04.20.537735
- [Background] Chen R, Del Rosario K, Lockman A, Boehm J, Bousquet Santos K, Siegel E, Berry Mendes W, Kubzansky LD. Effects of Induced Optimism on Subjective States, Physical Activity, and Stress Reactivity. J Posit Psychol. 2023;18(4):592-605. doi: 10.1080/17439760.2022.2070529. Epub 2022 May 8. PMID 37378047
- [Background] 4. Burke, K. L., Barry Joyner, A., Czech, D. R., & Wilson, M. J. (1989). An Investigation of Concurrent Validity between Two Optimism/Pessimism Questionnaires: The Life Orientation Test-Revised and the Optimisn essimism Scale. Marshall and Lang.
- [Background] Brown SD, Unger Hu KA, Mevi AA, Hedderson MM, Shan J, Quesenberry CP, Ferrara A. The multigroup ethnic identity measure-revised: measurement invariance across racial and ethnic groups. J Couns Psychol. 2014 Jan;61(1):154-161. doi: 10.1037/a0034749. Epub 2013 Nov 4. PMID 24188656
- [Background] 2. Bollwerk, M., Wetzel, E., Schlipphak, B., & Back, M. D. (2024). Who feels marginalized? A latent class analysis of perceived societal marginalization. Group Processes and Intergroup Relations, 27(3), 597-618. https://doi.org/10.1177/13684302231182924
- [Background] Bollwerk, M., Schlipphak, B., & Back, M. D. (2022). Development and Validation of the Perceived Societal Marginalization Scale. European Journal of Psychological Assessment, 38(2), 137-149. https://doi.org/10.1027/1015-5759/a000651